CLINICAL TRIAL: NCT05930808
Title: A Randomized, Open-label, 2-way-crossover Study Assessing the Bioequivalence Between Single Doses of 5 mg Concor® Tablets (Manufactured by Merck/China Nantong) and 5 mg Concor® Tablets (Manufactured by Merck/Germany Darmstadt) in Chinese Healthy Participants Under Fed or Fasted Conditions
Brief Title: Concor® Bioequivalence Study in Chinese Participants (Darmstadt-Nantong)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200006_0131
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Bisoprolol; Clinical equivalence; Pharmacokinetic
MeSH Terms: interventions — Bisoprolol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First Test Concor (Fasted), Then Reference Concor (Fasted) (Experimental): Participants will receive a single oral dose of Test Concor tablet on Day 1 in treatment period 1 followed by single oral dose of reference Concor tablet on Day 8 in treatment period 2 under fasted condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: First Test Concor (Fasted)
- First Reference Concor (Fasted), Then Test Concor (Fasted) (Experimental): Participants will receive a single oral dose of Reference Concor tablet on Day 1 in treatment period 1 followed by single oral dose of Test Concor tablet on day 8 in treatment period 2 under fasted condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: First Reference Concor (Fasted)
- First Test Concor (Fed), Then Reference Concor (Fed) (Experimental): Participants will receive a single oral dose of Test Concor tablet on Day 1 in treatment period 1 followed by a single oral dose of Reference Concor tablet on Day 8 in treatment period 2 under fed condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: First Test Concor (Fed)
- First Reference Concor (Fed), Then Test Concor (Fed) (Experimental): Participants will receive a single oral dose of Reference Concor tablet on Day 1 in treatment period 1 followed by a single oral dose of Test Concor tablet on Day 8 in treatment period 2 under fed condition. There will be separate washout period of 7 days between each treatment period.
  Interventions: Drug: First Reference Concor (Fed)

INTERVENTIONS:
Drug: First Test Concor (Fasted) — Participants will receive single oral dose of Test Concor tablet under fasted or fed condition.
  Other Names: Bisoprolol
  Arms: First Test Concor (Fasted), Then Reference Concor (Fasted)
Drug: First Reference Concor (Fasted) — Participants will receive single oral dose of Reference Concor tablet under fasted or fed condition
  Other Names: Bisoprolol
  Arms: First Reference Concor (Fasted), Then Test Concor (Fasted)
Drug: First Test Concor (Fed) — Participants will receive single oral dose of Test Concor tablet under fasted or fed condition.
  Other Names: Bisoprolol
  Arms: First Test Concor (Fed), Then Reference Concor (Fed)
Drug: First Reference Concor (Fed) — Participants will receive single oral dose of Reference Concor tablet under fasted or fed condition.
  Other Names: Bisoprolol
  Arms: First Reference Concor (Fed), Then Test Concor (Fed)

SUMMARY:
The purpose of this study is to assess is the bioequivalence (BE) of Concor 5 milligram (mg) tablets manufactured by Merck/China Nantong (test product) and Concor 5 mg tablets manufactured by Merck/Germany Darmstadt (reference product) in Chinese healthy participants under fed or fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests and cardiac monitoring
* Participant must have a body weight within 50-90 kilogram (kg) and body mass index (BMI) within the range 19-26 kilogram per meter square (kg/m2) (inclusive)
* Participant must have negative screen for alcohol and drugs of abuse at screening and on admission
* Both male and female participants. The Investigator confirms that each participant agrees to use appropriate contraception and barriers, if applicable
* Participant must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participant must not have any condition, including any uncontrolled disease state, that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Participant should not have positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, and treponema pallidum antibodies
* Participant must not have received any prescription or non-prescription medication within 28 days before the first study intervention administration, including multivitamins and herbal products (example, St John's Wort, or traditional Chinese medicines)
* Participant must not have participation in a study trial within 90 days prior to first drug administration; Blood donation (equal or more than 400 milliliter [mL]) or significant blood loss within 90 days prior to first drug administration
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Plasma Concentrations of Drug Concor under Fasted and Fed condition | Pre-dose up to 48 hours post-dose on Day 1 and Day 8

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, AEs Leading to Death, and AEs Leading to Discontinuation | Baseline up to Day 30 (approximately 4 weeks)
Number of Participants with Abnormal Vital Signs, Laboratory Variables, 12-Lead Electrocardiogram (ECG) and Physical Examination | Baseline up to Day 30 (approximately 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Beijing Friendship Hospital, Capital Medical University-Drug Clinical Trial Organization Office, Beijing, China

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200006_0131
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html